CLINICAL TRIAL: NCT05232396
Title: A Multi-center, Randomized, Double-blind Phase Ib Clinical Study to Evaluate the Safety, Tolerability, PK/PD Characteristics and Preliminary Efficacy of IL-6R mAb Injection in Patients With Active Moderate-to-Severe Rheumatoid Arthritis.
Brief Title: Clinical Study of Single Dose IL-6R mAb Injection in RA Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing VDJBio Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HJG-KBJS6-WDJ-Ⅰb
Record Dates: First submitted 2021-11-25; First posted 2022-02-09 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IL-6R Monoclonal Antibody Injection 4mg/kg (Experimental): IL-6R Monoclonal Antibody Injection 4mg/kg, single dose usage
  Interventions: Biological: IL-6R Monoclonal Antibody Injection 4mg/kg
- IL-6R Monoclonal Antibody Injection 6mg/kg (Experimental): IL-6R Monoclonal Antibody Injection 6mg/kg, single dose usage
  Interventions: Biological: IL-6R Monoclonal Antibody Injection 6mg/kg
- IL-6R Monoclonal Antibody Injection 8mg/kg (Experimental): IL-6R Monoclonal Antibody Injection 8mg/kg, single dose usage
  Interventions: Biological: IL-6R Monoclonal Antibody Injection 8mg/kg
- Tocilizumab Injection 8mg/kg (Active Comparator): Tocilizumab Injection 8mg/kg，as active comparator, single dose usage.
  Interventions: Biological: Tocilizumab Injection 8mg/kg

INTERVENTIONS:
Biological: IL-6R Monoclonal Antibody Injection 4mg/kg — IL-6R Monoclonal Antibody Injection 4mg/kg i.v.,single use
  Arms: IL-6R Monoclonal Antibody Injection 4mg/kg
Biological: IL-6R Monoclonal Antibody Injection 6mg/kg — IL-6R Monoclonal Antibody Injection 6mg/kg i.v. , single use
  Arms: IL-6R Monoclonal Antibody Injection 6mg/kg
Biological: IL-6R Monoclonal Antibody Injection 8mg/kg — IL-6R Monoclonal Antibody Injection 8mg/kg i.v. , single use
  Arms: IL-6R Monoclonal Antibody Injection 8mg/kg
Biological: Tocilizumab Injection 8mg/kg — Tocilizumab Injection 8mg/kg i.v., single use
  Arms: Tocilizumab Injection 8mg/kg

SUMMARY:
This is a single-dose,multi-center, randomized, double-blind, positive-controlled and parallel group clinical study that aims to evaluate the safety,tolerability,PK/PD characteristics and Preliminary Efficacy of Recombinant Humanized IL-6R Monoclonal Antibody Injection in Patients With Active Moderate-to-Severe Rheumatoid Arthritis.

DETAILED DESCRIPTION:
This study is aim to evaluate the safety, tolerability, PK/PD characteristics, immunogenicity parameters and Preliminary Efficacy of Recombinant Humanized IL-6R Monoclonal Antibody Injection in Patients With Active Moderate-to-Severe Rheumatoid Arthritis. There are 4 dose groups and each group enrolls 10 patients: 4mg/kg(IL-6R mAb); 6mg/kg(IL-6R mAb); 8mg/kg(IL-6R mAb) and 8mg/kg(tocilizumab ).each patient receives a single intravenous(i.v.) dose. The infusion time is from 60 to 90 minutes (the speed can be adjusted appropriately if there are injection reactions).

ELIGIBILITY:
Inclusion Criteria:

1. Age at the time of screening is 18~70 years old (including boundary value), gender is not limited;
2. According to the standards revised by the American College of Rheumatology (ACR) in 1987, or the American College of Rheumatology/Europe Anti-Rheumatism Alliance (ACR/EULAR) 2010 classification criteria, patients diagnosed with adult RA and The history of RA is at least 6 months;
3. Patients with moderate to severe active RA at screening and baseline visit, defined as having at least 6/68 joints Tenderness or pain and swelling of at least 6/66 joints during exercise After major surgical treatment, for the screening of this study, joint tenderness count (TJC) and closed The joint swelling count (SJC) evaluation, this joint cannot be counted);
4. Erythrocyte sedimentation rate (ESR) ≥28mm/hour, or C-reactive protein ≥ 10mg/L;
5. Before screening, due to lack of efficacy or intolerance, poor response to MTX treatment;
6. Have received and tolerated at least 7.5mg/week MTX treatment for at least 12 weeks before screening, and within 4 weeks before screening The dose of MTX is stable within the range of ≥7.5mg/week and ≤20mg/week. This MTX dose is expected to remain stable during the study period It will only be adjusted for safety reasons;
7. If subjects are using non-steroidal anti-inflammatory drugs (NSAIDs) or other analgesics to treat RA, they must be stable before enrollment.

   Fixed-dose treatment for at least 2 weeks;
8. If the subject takes glucocorticoids orally, the dose must be stabilized at least 4 weeks before enrollment to be equivalent to ≤10mg Prednisone/day dose;
9. Subjects who receive non-disabled concomitant drug treatment for any reason must always be on a stable treatment plan, definition It is that no new drug has been taken or the dosage has been changed within 7 days or 5 half-lives (whichever is longer) before screening;
10. Sign the informed consent form voluntarily.

Exclusion Criteria:

1. Have used DMARDs other than MTX (including sulfasalazine, antimalarial drugs, penicillamine, Azathioprine, cyclosporine A, cyclophosphamide, etc.), botanical drugs (including tripterygium wilfordii, total glucosides of paeony, sinomenine, etc.), and Those who have received any viral vaccine (such as influenza vaccine) immunotherapy;
2. Those who have had major trauma or undergone major surgery within 4 weeks before screening, or plan to receive medical treatment within 2 months after randomization.

   Those who have undergone major surgery;
3. Those who have used intra-articular, intramuscular or intravenous corticosteroids within 6 weeks before screening;
4. Anuranofin, gold glucosinolate (gold for injection), gold thiomalate (gold for injection) have been used within 8 weeks before screening Or those immunized with oral polio vaccine;
5. Those who received flunomide treatment within 12 weeks before screening (if receiving standard cholestyramine elution treatment 4 weeks before screening) (Cholestyramine 8g orally, 3 times a day for 11 consecutive days), then the subject can be included];
6. Those who have intravenous injection of gamma globulin, plasma exchange or use prosorba column within 24 weeks before screening;
7. Anakinra and Etanercept were used within 4 weeks before screening; Adalimumab and Etanercept were used within 8 weeks before screening Fliximab; Golimumab and Certuzumab used within 10 weeks before screening; Abba within 12 weeks before screening Cipro; used denosumab within 21 weeks before screening; used rituximab within 26 weeks before screening;
8. Those who have used tocilizumab in the past;
9. Uncontrolled cardiovascular system, respiratory system, digestive system, endocrine system, blood as judged by the investigator System, nervous system or psychiatric disorder or any other serious and/or unstable disease or medical history, and the investigator agrees For these diseases or medical history, taking study drugs may bring risks or interfere with the interpretation of data;
10. People with autoimmune diseases other than RA, including but not limited to psoriatic arthritis (PsA), ankylosing spine Inflammation (AS), systemic lupus erythematosus (SLE) or Lyme disease;
11. New York Heart Association functional class IV;
12. Non-metastatic basal cell carcinoma that has been adequately treated or resected in patients with malignant tumors or a history of malignant tumors Or squamous cell carcinoma or cervical cancer in situ;
13. The 12-lead electrocardiogram (ECG) is abnormal at the time of screening, and the investigator or sponsor believes that the abnormality has clinical significance And it may bring unacceptable risks to patients participating in this study (for example, Fridericia corrected QT interval>500 msec);
14. Laboratory screening test values have any of the following specific abnormalities:

    AST or ALT>2 times ULN; Total bilirubin >=1.5 times ULN; Hemoglobin <80.0g/L; Total white blood cell count<3.5×109/L; Neutropenia (absolute neutrophil count <1.5×109/L); Lymphopenia (lymphocyte count<0.75×109/L); Thrombocytopenia (platelet count<80×109/L); Creatinine> upper limit of normal; Triglycerides>10mmol/L;
15. Those with a history of infection of the prosthesis and the prosthesis is still in place;
16. There is evidence of active tuberculosis (TB), or there has been evidence of active TB before and has not received appropriate documented treatment; those with hidden tuberculosis infection are defined as tuberculin skin test (PPD) induration greater than 5mm Or those who have a positive interferon-gamma release test (such as TSPOT) and have not been treated for preventive tuberculosis for 4 weeks;
17. Patients with clinically significant infections within 6 months before screening (for example, those who need hospitalization or parenteral antibacterial treatment or opportunistic infections) Person), or have more than 1 oral or genital herpes, or history of herpes zoster, history of disseminated herpes, researchers Any history of infection that is judged to be likely to worsen due to participation in the study by other means, or need antibacterial within 2 weeks after screening Any person with a history of infections treated;
18. Those who plan to vaccinate or take oral vaccines during the study treatment period or within 8 weeks after study completion/early withdrawal;
19. Those with a history of any lymphoproliferative disease, such as EBV-related lymphoproliferative disease, lymphoma, leukemia, History of myeloproliferative disease, multiple myeloma, or current signs and symptoms of lymphatic disease;
20. People with uncontrolled asthma, psoriasis or inflammatory bowel disease who need oral corticosteroids for treatment;
21. Used before screening or planned to use lymphocyte depleting agents/therapies, alkylating agents, total lymphatic irradiation during the study period Other treatment methods;
22. Immediate family members or those who have hereditary immunodeficiency diseases;
23. Those who have been allergic to human or murine monoclonal antibodies in the past;
24. Those who suffer from active fibromyalgia and will make it difficult for researchers to accurately evaluate the RA activity in this study;
25. Serum virology examination: hepatitis B virus surface antigen, hepatitis C virus antibody, syphilis specific antibody, human Immunodeficiency virus-like virus antibody test, any one of which is positive;
26. With a history of alcohol or drug abuse, except for those who have been completely abstinent for more than 6 months before enrollment;
27. Those who have participated in any other clinical trials within 3 months before screening (only participated in the screening of clinical trials without using Except for subjects of test drugs);
28. Pregnant women, lactating women, or women of childbearing age who have a positive pregnancy test result during screening; or Those who have a childbirth plan during the trial period and within 3 months after the end of the study are unwilling to take it during the trial period and within 3 months after the end of the study One or more physical contraceptive measures;
29. The investigator believes that it is not suitable to participate in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Safety as measured by patients with adverse events | First dose up to last follow-up visit(Day1-Day57)
  The number of occurrences and incidence are calculated
AUC from time 0 to the time of the last quantifiable concentration AUC0-tlast of IL-6R | First dose up to last follow-up visit（Day1-Day57）
  AUC from time 0 to the time of the last quantifiable concentration AUC0-tlast of IL-6R
Maximum observed plasma concentration (Cmax) | First dose up to last follow-up visit（Day1-Day57）
  Maximum observed plasma concentration (Cmax) of IL-6R

SECONDARY OUTCOMES:
ACR20 ACR 50 ACR 70 response rate | At the 4th and 8th week of medication
  The ACR20, ACR50 or ACR70 was achieved if there was at least a 20%, 50% or 70% improvement from baseline in swollen joint count 66 (SJC66) and tender joint count 68 (TJC68) and 3 or more of the 5 following assessments: participant's assessment of pain, GH, physician's global assessment of disease activity, participant's assessment of physical function and CRP
Clinical Disease Activity Index (CDAI) response rate | At the 4th and 8th week of medication
  CDAI improvement ≥50% or CDAI≤2.8
HAQ- DI | At the 4th and 8th week of medication
  Changes in health Assessment Questionnaire disability Index (HAQ-DI) from baseline
FACIT-F | At the 4th and 8th week of medication
  Chronic Disease Functional Assessment - Fatigue Scale (FACIT-F) score was relatively basic Line changes
Analysis of immunogenicity | From Day15-Day71 after administration
  The concentrations of anti-drug antibody (ADA) and neutralizing antibody (NAb) in serum were detected

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, M.D., Principal Investigator — Peking University People's Hospital; Yi Fang, PhD, Principal Investigator — Peking University People's Hospital
Locations (5):
- China (5):
  - Affiliated Hospital of Hebei University, Baoding
  - Peking University People's Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Pingxiang City People's Hospital, Pingxiang
  - Peking University Shenzhen Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No